CLINICAL TRIAL: NCT02834663
Title: Prospective, Single-center, Six-month Study of Intravitreal Ranibizumab for Macular Edema With Nonproliferative Diabetic Retinopathy: Effects on Microaneurysm Turnover and Non-perfused Retinal Area
Brief Title: Effects of Intravitreal Ranibizumab for Macular Edema With Nonproliferative Diabetic Retinopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wonkwang University Hospital (Other)
Collaborators: Novartis Korea Ltd. (Industry)
Responsible Party: Principal Investigator, Yun-Sik Yang, MD, PhD, Wonkwang University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CRFB002DKR03T
Record Dates: First submitted 2016-06-26; First posted 2016-07-15 (Estimated); Results first posted 2020-04-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Nonproliferative Diabetic Retinopathy
Keywords: Nonproliferative diabetic retinopathy, Microaneurysms
MeSH Terms: conditions — Microaneurysm | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lucentis (Experimental): Patients were administered 0.5-mg IVR injections monthly for 6 months.
  Interventions: Drug: Lucentis

INTERVENTIONS:
Drug: Lucentis — Local anesthesia with T-caine with Saline irrigation. Routine eye drap was done by potadine-cotton ball. Lucentis injected to vitreous cavity, finally dressing.
  Other Names: Intravitreal Lucentis injection

SUMMARY:
Title of study:

Effects of Ranibizumab to delay or regression non-proliferative diabetic retinopathy(NPDR) with DME assessed by microaneurysm changes: A pilot study Objectives Diabetic retinopathy (DR) is a major cause of visual impairment. Anti-vascular endothelial growth factors have demonstrated therapeutic benefits in diabetic macular edema (DME). We aimed to prospectively analyze the effects of early intensive treatment using intravitreal ranibizumab (IVR) injections in nonproliferative diabetic retinopathy patients with macular edema.

Primary objective:

To investigate other efficacy endpoints including other visual acuity, anatomical change in mild-to-moderate NPDR with DME after intravitreal Ranibizumab injection from baseline through 6 months after treatment.

Secondary objectives:

To compare microvascular changes assessed by microaneurysm counts and perifoveal non-perfusion area changes and safty in eyes of mild-to-moderate NPDR with DME after intravitreal Ranibizumab injection from baseline through 6 months after treatment.

DETAILED DESCRIPTION:
Title of study:

Effects of Ranibizumab to delay or regression non-proliferative diabetic retinopathy(NPDR) with DME assessed by microaneurysm changes: A pilot study

Study Rationale:

Diabetic retinopathy is the leading disease that causes acquired vision loss after 20 by making diabetic macular edema and neovascularization. In recent young generation, as prevalence of type 2 diabetes is growing, the burden of sight-threatening retinopathy is increasing on trend.1 Pathologically, angiogenesis is a main cause that destroys the structure of the eye and induces the visual function disorder as VEGF playing an important role in increasing the migration and proliferation of endothelial cells and increasing the permeability of the blood vessels.2,3 VEGF is made from the endothelial cells of retinal tissue, perivascular cells, pigment endothelial cells by hypoxia. And hypoxic condition of intraocular tissues is a key regulator of intra ocular angiogenesis by VEGF, the balance between VEGF and angiogenesis inhibitors determines the neovascular proliferation in diabetic retinopathy.4 VEGF is also inducing the expression of cell-to-cell contact molecule (intracellular adhesion molecule-1, ICM-1) and the adhesion of leukocytes to help the inflammatory response5, as mediator which destroys the blood retinal barrier, affecting the protein of tight junctions, making a microaneurysm and increasing permeability of capillary, that makes the liquid leakage and macular edema.5,6 Microanuerysm is the earliest clinical manifestations, the saccular local lesion that perivascular cells protruding in damaged areas on the capillary wall. According to Stitt AW et al9, diabetic microaneurysm is non-functioning extrusion of the vascular system from the deep part of inner retinal capillary plexus.

It is sometimes disappeared by being blocked with blood clots, on the other hand, new microanerysm is occurred in the other vascular bed structure.

Through these changes, the investigators know the course of a diabetic retinopathy and it is known that the generation rate of microaneurysm is associated with the clinically significant progression of macular edema (CSME) in mild-to-moderate nonproliferative diabetic retinopathy .10,11 In addition, the number of microanerysm is an important prognostic indicator which can estimate the progression or regression of diabetic retinopathy, as predicting whether becoming better or worse in diabetic retinopathy.12 Kohner and Sleightholm13 describe this concept at first time in 1986, its association with the number of microvascular flow and the severity of diabetic retinopathy. In recent years it is reported that measuring the number of microaneurysm and the turnover rate associated with the appearance or disappearance of microaneurysm, are predictors in progression of diabetic retinopathy and macular edema.14 To delay the progression of diabetic retinopathy and to improve macular edema, the laser photocoagulation have been the important role.15 Although the laser photocoagulation have had treatment effect in the diabetic retinopathy by reducing the amount of VEGF in micraneurysm and by degenerating the neovascularization after laser therapy, there was a problem that has many limitations - peripheral visual field defects, night blindness, progression of macular edema etc., and that the disease does not cured in a good time because of limits of laser therapy due to cataract, vitreous hemorrhage and turbidity. As an alternative method to solve these limitations, there is an anti-VEGF therapy.6 According to a previous study result, intraocular injection of Bevacizumab inhibits occurring of neovascularization by blocking the VEGF receptor .17 Recently, several studies have been reported that when injected intravitreal anti-VEGF, macular edema is improved and neovascularization is inhibited, by reducing the leakage of neovascularization.3 Especially, Leicht SF et al18 reported the number of microaneurysms and turnover rate in NPDR(non-proliferative diabetic retinopathy) patients injected with Ranibizumab. And the result showed entire number of the microaneurysms and turnover rate are decreased, which could be mean the regression of diabetic retinopathy and it could decide the therapeutic effect.

On this study, through the fluorescein fundus angiography, the average number of microaneurysms was significantly decreased after intravitreal injection of anti-VEGF therapy (p<0.05). The decrease of 35.70±24.79% in the treatment group was statistically higher than 13.95±38.21% in the control group of the fellow eye (p<0.05).

The result is found because decreased concentration of intravitreal VEGF inhibits the progression of diabetic retinopathy, such as endothelial cell proliferation and endothelial cell damage on retinal capillary and perivascular cells.

Sjølie AK et al12 reported up-regulation of VEGF occuring microaneurysms causes endothelial cell proliferation and inflammation and effusion reaction, so anti-VEGF is effective in early diabetic retinopathy. But there is less effectiveness in late diabetic retinopathy as it reaches the non-changing point. Also Kohner EM et al19 reported diabetic retinopathy lesions are reversible and could be delayed in early diabetic retinopathy.

So far, changes of microaneurysms in late diabetic retinopathy is uncertain, and if there would be a finding according to anti-VEGF therapy, the investigators could get a clue of surrogate marker which represents treatment results in diabetic retinopathy.

This study was designed to find the clinical evaluation and reduction rate through fluorescein angiography as microaneurysm examination tools to research NPDR with DME treatment results assessed by microaneurysm counts, timely monitored with anti-VEGF therapy.

Objectives To evaluate the effects of intravitreal Ranibizumab injection on microvascular changes in eyes of mild-to-moderate NPDR with DME.

Primary objective:

To investigate other efficacy endpoints including other visual acuity, anatomical change in mild-to-moderate NPDR with DME after intravitreal Ranibizumab injection from baseline through 6 months after treatment.

Secondary objectives:

To compare microvascular changes assessed by microaneurysm counts and perifoveal non-perfusion area changes and safty in eyes of mild-to-moderate NPDR with DME after intravitreal Ranibizumab injection from baseline through 6 months after treatment.

Primary and secondary endpoints:

Primary endpoint:

To compare other visual acuity, anatomical changes after intravitreal Ranibizumab injection from baseline through 6 months after treatment.

i) The changes in best corrected visual acuity (BCVA) using ETDRS chart. ii) The central macular thickness - Circle Diameters : 1 mm ETDRS by spectralis OCT ; Heidelberg Engineering.

Secondary endpoints:

To compare microaneurysmal changes and perifoveal non-perfusion area and safty after intravitreal Ranibizumab injection from baseline through 6 months after treatment.

i) The total number of microaneurysm by fundus photo using Retmarker DR(version 1.0.2) software.

ii) The microaneurysm formation rate : Number of new MAs detected/month. iii) The microaneurysm disappearance rate : Number of MAs that resolved/month. iv)The microaneurysm turnover. v) Perifoveal non-perfusion area in FAG (mm²) using ImageJ software (version 1.52a) by FAG image.

vi) Safety parameters : Systemic adverse events (MI, CVA, etc), Ocular adverse events (retinal detachment, RPE tear, endophthalmitis, uveitis, vitreous hemorrhage, subretinal hemorrhage, cataract , IOP elevation, etc).

Methodology:

single center, prospective, interventional, one arm, pilot study

Evaluation Participants will be evaluated with a full ocular examination at each visit (VA measurement, tonometry, slit lamp exam). Fluorescein angiography (FA) will be performed at baseline, at 3 months after baseline and at the last visit(6 months after baseline), and OCT will be performed monthly (baseline and 1, 2, 3, 4, 5, 6 months from baseline).

The MAs and perifoveal non-perfused areas in individual retinas were evaluated at 6 months using fundus photography and FA imaging. The Retmarker (version 1.0.2 by Retmarker Ltd, Coimbra, Portugal) software was used for automatic measurement and analysis of changes in number and extent of MAs on fundus photographs and to calculate the total number and turnover of MAs.

Perifoveal non-perfused area was estimated using the early FA image (from each of the three examinations) in which both the vascular arch and the non-perfused area were clearly visualized. Subsequently, the ImageJ software (version 1.25a 23/04/2018 by ImageJ, USA) was used for scaling each image to 200 µm and for equalizing the contrast and sensitivity of each picture to the maximum possible extent, by auto-adjustment of brightness and contrast. The raw red-green-blue (RGB) images were then converted to 8-bit images, with the threshold set for optimal visualization of the non-perfused area. The same threshold was applied to all images of the same patient.

Result analysis The investigators compare the differences between at baseline, at 3 month, and at 6 month. Statistical analyses will be performed using SPSS ver.18.0 (SPSS Inc., Chicago, Il, USA). Kolmogorov-Smirnov test was applied to test for normality of sample group data. the paired T-test was used for comparative statistical analysis of these parameters. (BCVA, CRT, total number of MAs, MA formation rate, MA disappearance rate, MA turnover, and perifoveal non-perfused area)

ELIGIBILITY:
Inclusion Criteria:

* Patients (Male & female) ≥40 years of age
* Type 2 DM
* Best corrected visual acuity ≥ 20/200 (Snellen equivalent using Early Treatment Diabetic Retinopathy Study chart)
* central retinal thickness of ≥300 µm on optical coherence tomography
* nonproliferative diabetic retinopathy (NPDR) with diabetic macular edema

Exclusion Criteria:

* proliferative diabetic retinopathy
* Vitreous hemorrhage
* previous history of vitreoretinal surgery, post-cataract operation status (≤4 months before participation in this study)
* prior treatment with anti-VEGF drugs, intraocular corticosteroids, and/or retinal laser application
* Uncontrolled hypertension.
* Uncontrolled glaucoma.
* If both eyes met the study inclusion criteria, the more severely affected eye was selected

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yunsik Yang, MD, Ph D, Study Chair — Department of Ophthalmology, Wonkwang University School of Medicine; Seungjoon Lee, MD, Ph D, Principal Investigator — Study Official Affiliation should have no more than 80 characters.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liinamaa MJ, Savolainen MJ. High vitreous concentration of vascular endothelial growth factor in diabetic patients with proliferative retinopathy using statins. Ann Med. 2008;40(3):209-14. doi: 10.1080/07853890701749209. PMID 18382886
- [Background] Noma H, Funatsu H, Yamasaki M, Tsukamoto H, Mimura T, Sone T, Hirayama T, Tamura H, Yamashita H, Minamoto A, Mishima HK. Aqueous humour levels of cytokines are correlated to vitreous levels and severity of macular oedema in branch retinal vein occlusion. Eye (Lond). 2008 Jan;22(1):42-8. doi: 10.1038/sj.eye.6702498. Epub 2006 Jul 7. PMID 16826241
- [Background] Crawford TN, Alfaro DV 3rd, Kerrison JB, Jablon EP. Diabetic retinopathy and angiogenesis. Curr Diabetes Rev. 2009 Feb;5(1):8-13. doi: 10.2174/157339909787314149. PMID 19199892
- [Background] Usui T, Ishida S, Yamashiro K, Kaji Y, Poulaki V, Moore J, Moore T, Amano S, Horikawa Y, Dartt D, Golding M, Shima DT, Adamis AP. VEGF164(165) as the pathological isoform: differential leukocyte and endothelial responses through VEGFR1 and VEGFR2. Invest Ophthalmol Vis Sci. 2004 Feb;45(2):368-74. doi: 10.1167/iovs.03-0106. PMID 14744874
- [Background] Hoeben A, Landuyt B, Highley MS, Wildiers H, Van Oosterom AT, De Bruijn EA. Vascular endothelial growth factor and angiogenesis. Pharmacol Rev. 2004 Dec;56(4):549-80. doi: 10.1124/pr.56.4.3. PMID 15602010
- [Background] Roy S, Ha J, Trudeau K, Beglova E. Vascular basement membrane thickening in diabetic retinopathy. Curr Eye Res. 2010 Dec;35(12):1045-56. doi: 10.3109/02713683.2010.514659. Epub 2010 Oct 7. PMID 20929292
- [Background] Hammes HP. Pericytes and the pathogenesis of diabetic retinopathy. Horm Metab Res. 2005 Apr;37 Suppl 1:39-43. doi: 10.1055/s-2005-861361. PMID 15918109
- [Background] Stitt AW, Gardiner TA, Archer DB. Histological and ultrastructural investigation of retinal microaneurysm development in diabetic patients. Br J Ophthalmol. 1995 Apr;79(4):362-7. doi: 10.1136/bjo.79.4.362. PMID 7742285
- [Background] Ribeiro ML, Nunes SG, Cunha-Vaz JG. Microaneurysm turnover at the macula predicts risk of development of clinically significant macular edema in persons with mild nonproliferative diabetic retinopathy. Diabetes Care. 2013 May;36(5):1254-9. doi: 10.2337/dc12-1491. Epub 2012 Nov 30. PMID 23204247
- [Background] Haritoglou C, Kernt M, Neubauer A, Gerss J, Oliveira CM, Kampik A, Ulbig M. Microaneurysm formation rate as a predictive marker for progression to clinically significant macular edema in nonproliferative diabetic retinopathy. Retina. 2014 Jan;34(1):157-64. doi: 10.1097/IAE.0b013e318295f6de. PMID 23792485
- [Background] Sjolie AK, Klein R, Porta M, Orchard T, Fuller J, Parving HH, Bilous R, Aldington S, Chaturvedi N. Retinal microaneurysm count predicts progression and regression of diabetic retinopathy. Post-hoc results from the DIRECT Programme. Diabet Med. 2011 Mar;28(3):345-51. doi: 10.1111/j.1464-5491.2010.03210.x. PMID 21309844
- [Background] Kohner EM, Sleightholm M. Does microaneurysm count reflect severity of early diabetic retinopathy? Ophthalmology. 1986 May;93(5):586-9. doi: 10.1016/s0161-6420(86)33692-3. PMID 3725317
- [Background] Nunes S, Pires I, Rosa A, Duarte L, Bernardes R, Cunha-Vaz J. Microaneurysm turnover is a biomarker for diabetic retinopathy progression to clinically significant macular edema: findings for type 2 diabetics with nonproliferative retinopathy. Ophthalmologica. 2009;223(5):292-7. doi: 10.1159/000213639. Epub 2009 Apr 16. PMID 19372723
- [Background] Photocoagulation treatment of proliferative diabetic retinopathy. Clinical application of Diabetic Retinopathy Study (DRS) findings, DRS Report Number 8. The Diabetic Retinopathy Study Research Group. Ophthalmology. 1981 Jul;88(7):583-600. PMID 7196564
- [Background] Ferrara N, Hillan KJ, Gerber HP, Novotny W. Discovery and development of bevacizumab, an anti-VEGF antibody for treating cancer. Nat Rev Drug Discov. 2004 May;3(5):391-400. doi: 10.1038/nrd1381. No abstract available. PMID 15136787
- [Background] Han XX, Guo CM, Li Y, Hui YN. Effects of bevacizumab on the neovascular membrane of proliferative diabetic retinopathy: reduction of endothelial cells and expressions of VEGF and HIF-1alpha. Mol Vis. 2012;18:1-9. Epub 2012 Jan 1. PMID 22232563
- [Background] Leicht SF, Kernt M, Neubauer A, Wolf A, Oliveira CM, Ulbig M, Haritoglou C. Microaneurysm turnover in diabetic retinopathy assessed by automated RetmarkerDR image analysis--potential role as biomarker of response to ranibizumab treatment. Ophthalmologica. 2014;231(4):198-203. doi: 10.1159/000357505. Epub 2014 Mar 19. PMID 24662930
- [Background] Kohner EM, Stratton IM, Aldington SJ, Turner RC, Matthews DR. Microaneurysms in the development of diabetic retinopathy (UKPDS 42). UK Prospective Diabetes Study Group. Diabetologia. 1999 Sep;42(9):1107-12. doi: 10.1007/s001250051278. PMID 10447523
- [Background] Horii T, Murakami T, Nishijima K, Sakamoto A, Ota M, Yoshimura N. Optical coherence tomographic characteristics of microaneurysms in diabetic retinopathy. Am J Ophthalmol. 2010 Dec;150(6):840-8. doi: 10.1016/j.ajo.2010.06.015. Epub 2010 Sep 19. PMID 20855054

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an interventional, prospective, single-center study conducted at Wonkwang University Hospital from August 2016 to February 2019. All patients included in the study provided signed, informed consent prior to enrollment.
Pre-assignment Details: previous history of vitreoretinal surgery, post-cataract operation status (≤4 months before participation in this study), uncontrolled hypertension, or glaucoma were excluded from the study.
Units Other Than Participants: eyes
Groups:
- Lucentis(Ranivizumab): 25 eyes of 25 type 2 diabetes mellitus patients with macular edema were included between August 2016 and February 2019. For 6 months, patients were administered 0.5-mg intra-vitreal Lucentis(Ranibizumab) injections monthly.
Period: Overall Study
Arm/Group | Lucentis(Ranivizumab)
Started | 25; 25 eyes (Unit means the eye. One eye was included per patient)
Completed | 25; 25 eyes (Unit means the eye. One eye was included per patient)
Not Completed | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: Totally, 25 eyes of 25 patients (13 males, 12 females, mean age 63.80±11.45 years; range: 41-80 years) were included in the study
Groups:
- Baseline Characteristics: Totally, 25 eyes of 25 patients (13 males, 12 females, mean age 63.80±11.45 years; range: 41-80 years) were included in the study
Arm/Group | Baseline Characteristics
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.80 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 25
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Duration of Diabetes Mellitus(DM) (year) [Mean (Standard Deviation); unit: years] | 12.04 (7.475)
HbA1c(%) [Mean (Standard Deviation); unit: %] | 8.27 (2.11)
BCVA (ETDRS letters) [Mean (Standard Deviation); unit: ETDRS letters] — ETDRS charts present a series of five letters of equal difficulty on each row for a total of 14 lines (70 letters). An ETDRS letter score can be calculated as follows: when 20 or more letters are read correctly at 4.0 m, the visual acuity letter score is equal to the total number of letters read correctly at 4.0 m plus 30. If fewer than 20 letters are read correctly at 4.0 m, the visual acuity letter score is equal to the total number of letters read correctly at 4.0 m plus the total number of letters read correctly at 1.0 m in the first six lines.
  ETDRS letters | 67.60 (3.29)
CRT (um) [Mean (Standard Deviation); unit: um] — Central retinal thickness (CRT) was measured using optical coherence tomography
  um | 479.12 (16.66)
Total microaneurysms (number) [Mean (Standard Deviation); unit: microaneurysms] | 5.68 (3.41)
Microaneurysm-turnover [Mean (Standard Deviation); unit: microaneurysms/month] — MA turnover was calculated by adding the MA formation rate (number of new MAs detected/month) to the MA disappearance rate (number of MAs that resolved/month)
  microaneurysms/month | 6.88 (3.83)
Perifoveal non-perfused area (mm^2) [Mean (Standard Deviation); unit: mm^2] | 2.517 (0.456)

OUTCOME MEASURES:

1. Primary Outcome: The Best Corrected Visual Acuity (BCVA)
Description: BCVA was performed using the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at baseline and 6 months. The BCVA compare the degree of improvement or worsening of vision at baseline and 6 months. (value at 6 months minus value at baseline)
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: letters
Groups:
- BCVA Baseline: Before the treatment regimen, assessment of BCVA using the ETDRS charts.
- BCVA Resulte: After completion of the treatment regimen during 6 months, assessment of BCVA using the ETDRS charts.
Arm/Group | BCVA Baseline | BCVA Resulte
Number analyzed (Participants) | 25 | 25
letters | 67.6 (3.29) | 76.36 (1.61)
Statistical Analysis 1: Comparison: BCVA Baseline vs BCVA Resulte; Patients were evaluated for changes in BCVA of the treated eye, from the start of the study till 6 months, until trial completion. After administration of each injection, measurements of BCVA were compared to their respective baseline results. The paired t-test and repeated measures ANOVA was performed for comparative analysis, as all showed normality; Test type: Superiority; p < 0.0001, t-test, 2 sided — The threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = -8.760, 95% CI 2-sided [-13.928 to -3.592], Standard Deviation 12.521

2. Primary Outcome: Central Macular Thickness(CMT)
Description: CRT was performed using OCT at each visit. The OCT measured at each visit was analyzed statistically. the CMT compare the degree of improvement or worsening of vision at baseline and 6 months. (value at 6 months minus value at baseline)
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: um
Groups:
- CRT Baseline: Before the treatment regimen, assessment of CRT using the OCT.
- CRT Resulte: After the treatment regimen during 6 months, assessment of CRT using the OCT.
Arm/Group | CRT Baseline | CRT Resulte
Number analyzed (Participants) | 25 | 25
um | 479.12 (16.66) | 369.12 (13.02)
Statistical Analysis 1: Comparison: CRT Baseline vs CRT Resulte; Test type: Superiority; p = 0.0001, t-test, 2 sided — The threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = 110, 95% CI 2-sided [82.790 to 137.210], Standard Deviation 65.919

3. Secondary Outcome: The Total Number of Microaneurysm
Description: The number of MAs in individual retinas were evaluated during 6 months using fundus photography and FA imaging. The Retmarker software was used for automatic measurement and analysis of changes in number and extent of MAs on fundus photographs and to calculate the total number and turnover of MAs. Changes in MAs were analyzed statistically. the total number of MAs compare the degree of improvement or worsening of vision at baseline and 6 months. (value at 6 months minus value at baseline)
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: microaneurysms
Groups:
- Total MA Baseline: The number of MAs in individual retinas were evaluated at first visit using fundus photography and FA imaging. The Retmarker software was used for automatic measurement and analysis of changes in number and extent of MAs on fundus photographs and to calculate the total number and turnover of MAs.
- Total MA Resulte: The number of MAs in individual retinas were evaluated during 6 months using fundus photography and FA imaging. The Retmarker software was used for automatic measurement and analysis of changes in number and extent of MAs on fundus photographs and to calculate the total number and turnover of MAs.
Arm/Group | Total MA Baseline | Total MA Resulte
Number analyzed (Participants) | 25 | 25
microaneurysms | 5.68 (3.41) | 1.60 (1.73)
Statistical Analysis 1: Comparison: Total MA Baseline vs Total MA Resulte; Test type: Superiority; p = 0.001, t-test, 2 sided — The threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = 3.920, 95% CI 2-sided [1.884 to 5.956], Standard Deviation 4.932

4. Secondary Outcome: The Microaneurysm Formation Rate
Description: number of new MAs detected/month The MAs in individual retinas were evaluated at 6 months using fundus photography. The Retmarker (version 1.0.2 by Retmarker Ltd, Coimbra, Portugal) software was used for automatic measurement and analysis of changes in number and extent of MAs on fundus photographs and to calculate the total number and turnover of MAs. MA turnover was calculated by adding the MA formation rate (number of new MAs detected/month) to the MA disappearance rate (number of MAs that resolved/month). The microaneurysm formation rate compare the degree of improvement or worsening of vision at baseline and 6 months. (value at 6 months minus value at baseline)
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: microaneurysms/month
Groups:
- The MA Formation Rate Baseline: The Retmarker software was used for automatic measurement and analysis of MA formation at first visit.
- The MA Formation Rate Resulte: The Retmarker software was used for automatic measurement and analysis of MA formation during monthly 6 months
Arm/Group | The MA Formation Rate Baseline | The MA Formation Rate Resulte
Number analyzed (Participants) | 25 | 25
microaneurysms/month | 2.48 (1.98) | 0.96 (1.02)
Statistical Analysis 1: Comparison: The MA Formation Rate Baseline vs The MA Formation Rate Resulte; Test type: Superiority; p = 0.0001, t-test, 2 sided — The threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = 2.23, 95% CI 2-sided [1.30 to 3.15], Standard Deviation 2.24

5. Secondary Outcome: The Microaneurysm Disappearance Rate
Description: Number of MAs that resolved/month The MAs in individual retinas were evaluated at 6 months using fundus photography. The Retmarker (version 1.0.2 by Retmarker Ltd, Coimbra, Portugal) software was used for automatic measurement and analysis of changes in number and extent of MAs on fundus photographs and to calculate the total number and turnover of MAs. MA turnover was calculated by adding the MA formation rate (number of new MAs detected/month) to the MA disappearance rate (number of MAs that resolved/month). The microaneurysm disappearance rate compare the degree of improvement or worsening of vision at baseline and 6 months. (value at 6 months minus value at baseline)
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: microaneurysms/month
Groups:
- The MA Disappearance Rate Baseline: The Retmarker software was used for automatic measurement and analysis of MA disappearance at first visit.
- The MA Disappearance Rate Resulte: The Retmarker software was used for automatic measurement and analysis of MA disappearance during monthly 6 months.
Arm/Group | The MA Disappearance Rate Baseline | The MA Disappearance Rate Resulte
Number analyzed (Participants) | 25 | 25
microaneurysms/month | 4.40 (2.66) | 0.96 (1.09)
Statistical Analysis 1: Comparison: The MA Disappearance Rate Baseline vs The MA Disappearance Rate Resulte; Test type: Superiority; p = 0.0001, t-test, 2 sided — The threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = 5.64, 95% CI 2-sided [2.67 to 8.62], Standard Deviation 7.21

6. Secondary Outcome: The Microaneurysm Turnover
Description: The microaneurysm formation rate + The microaneurysm disappearance rate The MAs in individual retinas were evaluated at 6 months using fundus photography. The Retmarker (version 1.0.2 by Retmarker Ltd, Coimbra, Portugal) software was used for automatic measurement and analysis of changes in number and extent of MAs on fundus photographs and to calculate the total number and turnover of MAs. MA turnover was calculated by adding the MA formation rate (number of new MAs detected/month) to the MA disappearance rate (number of MAs that resolved/month). The microaneurysm turnover compare the degree of improvement or worsening of vision at baseline and 6 months. (value at 6 months minus value at baseline)
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: microaneurysms/month
Groups:
- The Microaneurysm Turnover Baseline: The Retmarker software was used for automatic measurement and analysis of MA turnover at first visit.
- The Microaneurysm Turnover Results: The Retmarker software was used for automatic measurement and analysis of MA turnover during monthly 6 months.
Arm/Group | The Microaneurysm Turnover Baseline | The Microaneurysm Turnover Results
Number analyzed (Participants) | 25 | 25
microaneurysms/month | 6.88 (3.83) | 1.92 (1.75)
Statistical Analysis 1: Comparison: The Microaneurysm Turnover Baseline vs The Microaneurysm Turnover Results; Test type: Superiority; p = 0.0001, t-test, 2 sided — The threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = 5.64, 95% CI 2-sided [2.67 to 8.62], Standard Deviation 7.21

7. Secondary Outcome: Perifoveal Non-perfusion Area in FAG (mm²)
Description: Using ImageJ software (version 1.52a) by FAG image. The Perifoveal non-perfusion area in FAG compare the degree of improvement or worsening of vision at baseline and 6 months. (value at 6 months minus value at baseline)
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mm2
Groups:
- Perifoveal Non-perfusion Area Baseline: The perifoveal non-perfused areas in individual retinas were evaluated at first visit using fundus photography and FA imaging. The Retmarker software was used for automatic measurement and analysis of changes in number and extent of MAs on fundus photographs and to calculate the total number and turnover of MAs
- Perifoveal Non-perfusion Area Results: The perifoveal non-perfused areas in individual retinas were evaluated during monthly 6 months using fundus photography and FA imaging. The Retmarker software was used for automatic measurement and analysis of changes in number and extent of MAs on fundus photographs and to calculate the total number and turnover of MAs
Arm/Group | Perifoveal Non-perfusion Area Baseline | Perifoveal Non-perfusion Area Results
Number analyzed (Participants) | 25 | 25
mm2 | 2.517 (0.456) | 2.495 (0.293)
Statistical Analysis 1: Comparison: Perifoveal Non-perfusion Area Baseline vs Perifoveal Non-perfusion Area Results; Test type: Superiority; p = 0.221, t-test, 2 sided — The threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = 0.021, 95% CI 2-sided [-0.751 to 0.795], Standard Deviation 1.87

8. Secondary Outcome: Safety Parameters
Description: Systemic adverse events (MI, CVA, etc), Ocular adverse events (retinal detachment, RPE tear, endophthalmitis, uveitis, vitreous hemorrhage, subretinal hemorrhage, cataract , IOP elevation, etc) at baseline and each visit.
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Safety Parameters Results: Complications and adverse events on patients were evaluated.
Arm/Group | Safety Parameters Results
Number analyzed (Participants) | 25
Participants | 0

ADVERSE EVENTS:
Time Frame: Twenty-five eyes of 25 type 2 diabetes mellitus patients with DME were included between August 2016 and February 2019. For 6 months, patients were administered 0.5-mg IVR injections monthly.
Description: Ocular evaluation, including best-corrected visual acuity (BCVA; using the Early Treatment Diabetic Retinopathy Study chart), central retinal thickness (CRT; using optical coherence tomography), fundus photography, and fluorescein angiography, was performed for all participants. Results obtained at baseline were compared to those observed after 6 months.
Groups:
- Adverse Event: Systemic adverse events (MI, CVA, etc), Ocular adverse events (retinal detachment, RPE tear, endophthalmitis, uveitis, vitreous hemorrhage, subretinal hemorrhage, cataract , IOP elevation, etc) on patients were evaluated.
Arm/Group | Adverse Event
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT02834663/Prot_SAP_000.pdf
  • Informed Consent Form (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT02834663/ICF_001.pdf